CLINICAL TRIAL: NCT05651542
Title: A Comprehensive Self-Management Intervention for Individuals With Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Kendra Kamp, Assistant Professor, Biobehavioral Nursing & Health Informatics, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY00015210; 1K23NR020044-01A1 (NIH)
Record Dates: First submitted 2022-12-05; First posted 2022-12-15 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Inflammatory Bowel Diseases; Ulcerative Colitis; Crohn Disease
Keywords: IBD; UC; CD
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive Self-Management (Experimental): The 8 week intervention is delivered online with a brief weekly check-in with a registered nurse.
  Interventions: Behavioral: Comprehensive Self-Management Intervention
- Usual care group (Other): The control group will receive standard care without the comprehensive self-management intervention.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Comprehensive Self-Management Intervention — In addition to standard care, participants receive content on self-management which includes cognitive behavioral therapy, relaxation, and diet. Weekly phone calls provide support for achieving the sessions goals.
  Arms: Comprehensive Self-Management
Other: Control — The control group will receive standard care.
  Arms: Usual care group

SUMMARY:
This study aims to test the feasibility, acceptability, and preliminary efficacy of a comprehensive self-management (CSM) intervention for people with inflammatory bowel disease (IBD). The CSM-IBD intervention is an adaption of the CSM intervention initially developed for individuals with irritable bowel syndrome. The intervention has eight sessions which cover an introduction to IBD, symptom tracking, cognitive behavioral strategies, relaxation, sleep, diet, and pain management.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare provider diagnosis of inflammatory bowel disease
* Report current symptoms
* Able to read and write in English

Exclusion Criteria:

* Live outside of Washington state
* Bowel-related surgery within the past month

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Recruitment feasibility | From screening to enrollment
  Percentage comprised of number of participants enrolled divided by the number of participants approached.
Intervention feasibility | 3 months
  Measured with the Feasibility of Intervention Measure (FIM) in which participants respond to four questions on a 5-point Likert scale from completely disagree (1) to completely agree (5).
Acceptability | 6 months
  A semi-structured interview guide will be used to assess acceptability of study procedures as well as acceptability and satisfaction with the intervention.

SECONDARY OUTCOMES:
Change in Quality of Life | Baseline, 3 months, 6 months
  Short Inflammatory Bowel Disease Questionnaire is a 10-item questionnaire which evaluates quality of life. Participants respond on a 7-item Likert scale from all the time to none of the time. Total score range: 10 to 70.
Change in Symptoms | Baseline, 3 months, 6 months
  Symptoms are measured using a numeric rating scale where participants report the severity of the symptom from not present (0) to worst possible (10). Symptoms include: abdominal pain, anxiety, bloating, constipation, depressed, diarrhea, fatigue/tiredness, passing gas, sleepiness during the day, stress, and urgency.

OTHER OUTCOMES:
Self-Efficacy for Managing Chronic Disease | Baseline, 3 months, 6 months
  a 6-item self-report scale. Participants report ranging from not at all confident to totally confident.
Index of Self-Regulation | Baseline, 3 months, 6 months
  a 9-item scale to measure individual's level of self-regulation
Patient Activation Measure | Baseline, 3 months, 6 months
  a 13-item scale which assess patient's beliefs, knowledge and confidence in managing their health
Fecal Calprotectin | Baseline, 3 months
  Level of fecal calprotectin assessed using ELISA.
Gut Microbiome | Baseline, 3 months
  Fecal microbial communities characterized using 16S rRNA gene sequencing on the Illumina MiniSeq platform (Illumina, Inc. Albany, New York)

CONTACTS AND LOCATIONS:
Overall Officials: Kendra Kamp, PHD, RN, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391
- [Derived] Kamp K, Clark-Snustad K, Yoo L, Winders S, Cain K, Levy RL, Dey N, Lee S, Keefer L, Heitkemper M. A Comprehensive Self-Management Intervention for Inflammatory Bowel Disease (CSM-IBD): Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2023 Jun 7;12:e46307. doi: 10.2196/46307. PMID 37285195

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT05651542/Prot_SAP_000.pdf